CLINICAL TRIAL: NCT03774056
Title: A Phase I Study Evaluating Tolerability, Pharmacokinetics, and Preliminary Efficacy of HC-1119 in Patients With Metastatic Castration-Resistant Prostate Cancer.
Brief Title: A Study Evaluating Tolerability, Pharmacokinetics, and Preliminary Efficacy of HC-1119 in Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC-1119-01
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose group (Experimental): Drug name L:HC-1119 Dosage: 40 mg, 80 mg, 160 mg, and 200 mg
  Interventions: Drug: HC-1119

INTERVENTIONS:
Drug: HC-1119 — oral

SUMMARY:
This is a phase I study evaluating tolerability, pharmacokinetics, and preliminary efficacy of HC-1119 in patients with metastatic castration-resistant prostate cancer. The study objective is to study the tolerability, safety, and dose-limiting toxicities (DLT) of HC-1119 in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria (those who meet all of the following are eligible):

1. Voluntarily participated in the study, with understanding of relevant study procedures and signed informed consent form;
2. Male , ≥18 years old;
3. With histologically or cytologically confirmed prostate cancer, without neuroendocrine carcinoma or ductal adenocarcinoma;
4. With evidence of metastatic disease (such as bone scan and CT/MRI results);
5. Patients with relapsed, refractory, or progressive disease despite castration (surgery or chemical) or combined androgen deprivation therapy (Progressive disease is defined as 1 or more of the following 3 criteria: Serum PSA progression: A minimum of 3 rising PSA values with an interval of at least 1 week between determinations, resulting in a final value higher than 50% of the minimum, with a starting PSA value > 2 ng/ml; Soft tissue disease progression as defined by RECIST 1.1; Bone disease progression defined by PCWG2 with 2 or more new metastatic lesions on bone scan);
6. Castrate levels of testosterone (< 50 ng/dl) at screening;
7. Bilateral orchiectomy or ongoing androgen deprivation therapy with effective GnRH analogues;
8. Estimated life expectancy > 6 months;
9. ECOG performance status ≤ 1;
10. Laboratory tests must meet the following criteria:

    1. Routine Blood Test: hemoglobin (Hb) ≥ 90 g/L (no blood transfusion within the last 14 days); absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count (PLT) ≥ 80 x 109/L;
    2. Blood Biochemistry: creatinine (Cr) ≤ 2 x upper limit of normal (ULN), or Cr > 2 x ULN but the calculated CrCl ≥ 60 mL/min; bilirubin (BIL) ≤ 2 x ULN; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x ULN (or ≤ 5.0 x ULN for patients with liver metastases);
    3. Coagulation: INR < 1.5.

Exclusion Criteria (those who meet any one of the following are ineligible):

1. Ongoing toxicity ( ≥ Grade 2 toxicity) from previous treatments;
2. Clinically significant GI dysfunction which may affect the intake, transport, or absorption of drug (such as inability to swallow, chronic diarrhea, and bowel obstruction, etc.), or patients with complete gastrectomy;
3. History of allergies, or known hypersensitivity to components of the investigational drug;
4. Brain metastases;
5. Other malignancies within the last 5 years (except for curatively treated non-melanoma skin cancer);
6. History of organ transplants
7. HIV seropositive;
8. Past medical history of seizures or serious CNS diseases;
9. History of unexplained coma;
10. Family history of seizures;
11. History of traumatic brain injury;
12. History of medication or drug abuse;
13. Patients with severe cardiovascular diseases, including those with myocardial infarction, arterial thrombosis, unstable angina, or clinical symptomatic heart failure within the past 6 months;
14. Uncontrolled hypertension (systolic ≥ 160 mmHg or diastolic ≥ 100 mmHg). Patients with a history of hypertension is eligible if his blood pressure is controlled with antihypertensives;
15. Medications that lower the seizure threshold must be used during the study;
16. Treatment with 5α-reductase inhibitors (finasteride, dutasteride), estrogen, or cyproterone within the past 4 weeks;
17. Treatment with ketoconazole within the past 4 weeks;
18. Previously treated with investigational or approved medications that inhibit testosterone synthesis (such as abiraterone acetate, TAK-683, and TAK-448) or target testosterone receptors (such as enzalutamide, SHR3680, proxalutamide, and ARN509);
19. Participated in other clinical trials within 1 month prior to enrollment;
20. Subjects is determined by the investigator to be unsuitable for this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities(DLT) | From the first dose of the study to the 12th week after dose
  Safety measures
Number of patients with adverse events | From the first dose of the study to the 12th week after dose
  Safety measures

SECONDARY OUTCOMES:
Maximum drug concentration(Cmax) | From the first dose of the study to the 12th week after dose
  Single-dose and repeated-dose
Time of maximum drug concentration(Tmax) | From the first dose of the study to the 12th week after dose
  Single-dose and repeated-dose
Area under curve from time 0 to 24h (AUC0-24h) | From the first dose of the study to the 12th week after dose
  Single-dose and repeated-dose
Maximal PSA Response Rate | From the first dose of the study to the 12th week after dose
  Percentage of patients with > 50% decrease in PSA levels from baseline during the 12-week treatment period
Response rate of prostate specific antigen (PSA) | From the first dose of the study to the 12th week after dose
  Percentage of patients with > 50% decrease in PSA levels from baseline at weeks 6, 8, 10, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, professor, Principal Investigator — West China Hospital; Li Zheng, professor, Principal Investigator — West China Hospital
Locations (1):
- Hinova Pharmaceuticals Inc., Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li X, Cheng K, Li X, Zhou Y, Liu J, Zeng H, Chen Y, Liu X, Zhang Y, Wang Y, Bi F, Zheng L. Phase I clinical trial of HC-1119: A deuterated form of enzalutamide. Int J Cancer. 2021 Oct 1;149(7):1473-1482. doi: 10.1002/ijc.33706. Epub 2021 Jul 7. PMID 34109624